CLINICAL TRIAL: NCT02813356
Title: United States Post-Marketing Observational Cardiovascular Safety Study in Patients Taking Naloxegol
Brief Title: Naloxegol US PMR CV Safety.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Valinor Pharma LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: D3820R00008; EUPAS18201 (Registry Identifier: ENCePP)
Record Dates: First submitted 2016-06-07; First posted 2016-06-27 (Estimated); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Opioid Induced Constipation
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — naloxegol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (2):
- naloxegol: patients exposed to naloxegol
  Interventions: Drug: naloxegol
- non-PAMORA: patients exposed to non-peripherally acting mu-opioid antagonist
  Interventions: Drug: non-PAMORA

INTERVENTIONS:
Drug: naloxegol — non-interventional study where naloxegol is prescribed during normal clinical practice
  Groups: naloxegol
Drug: non-PAMORA — non-interventional study where patients are exposed to non-peripherally acting mu-opioid antagonists during the normal course of clinical practice
  Groups: non-PAMORA

SUMMARY:
The overall research goal for this study is to provide additional data to characterize the safety of naloxegol in patients aged 18 years and older who do not have a diagnosis of cancer and who are treated with opioids chronically

DETAILED DESCRIPTION:
The primary objective is to assess the overall risk of major adverse cardiovascular events (MACE) among naloxegol-treated patients compared to that among patients on prescription non-peripherally acting mu-opioid antagonist (PAMORA) opioid induced constipation (OIC) treatment. The corresponding analysis is of a new-user cohort study that captures the occurrence of MACE in persons receiving naloxegol or comparison medications. The study takes place in actual-use settings in the US in which existing electronic data captures patient diagnoses, health care, and treatment. The occurrence of MACE in naloxegol-treated patients will be compared to the occurrence of MACE in medically-similar new users of other prescription-only treatments for OIC in the same settings, with both naloxegol-treated and comparison medication-treated patients being followed for as long as they continue on therapy.

In further pursuit of the primary objective, there will be a self-controlled study that follows all members of the new-user cohorts, including both new naloxegol users and new users of comparator products, for as long as data are available as the patients may go on or off treatment. A self-controlled study offers a complementary approach to the statistical control for the possible confounding effects of personal characteristics. Using the same data sources, this self-controlled design follows individuals from the time they finish their first course of treatment as new users for as long as the study continues. Patient treatment statuses are continuously updated since the treatment choices exercised by patients and their caregivers create extended periods of study time on and off naloxegol and possibly on and off other therapies for OIC. Comparisons of the occurrence of MACE occur within individuals and so are unaffected by differences between individuals, as in a crossover trial.

The first secondary objective is to assess the potential confounding effects of lifestyle risk factors on relative risk of MACE among naloxegol-treated patients compared with that among patients on other prescription non-PAMORA OIC treatment. The corresponding analysis is of a case-control study nested within the primary study population. All of the MACE "cases" will be matched to other members of the cohorts ("controls"). In cases and controls, the outpatient medical record will be abstracted for information on lifestyle risk factors. The case-control analysis will provide information on the presence and effect of lifestyle confounding factors that may be identifiable only by chart review.

Further secondary analyses will investigate the relative risks analyzed under an intent-to-treat paradigm over fixed time periods of membership in the naloxegol and comparator cohorts, relative risks for specific components of MACE, relative risks associated with new oral PAMORA agents other than naloxegol (non-naloxegol oral PAMORAs [NNPAMORAs]) that may come onto the US market during the course of the study, and an exploration of the possible variations in risk associated with variations in the dose and timing of naloxegol dispensing in the case-control study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient receives a new dispensing of naloxegol, lubiprostone/linaclotide, or an oral NNPAMORA. A new dispensing is one that occurs with no dispensing for the same drug having occurred in the preceding 182 days. A patient only qualifies once under this criterion for any drug.
2. Patients 18 years of age or older at the index date
3. Continuous availability of data for at least 183 days immediately before and including the index date
4. 90 days of opioid dispensed in the 183 days before and including the index date of which at least 30 days of opioid dispensed at at least 30 MEQ/day in the 60 days before and including index date
5. Current users of a dispensed opioid, meaning that the interval between index study drug dispensing and at least 1 prior opioid dispensing is less than the days supply associated with the opioid dispensing

Exclusion Criteria:

1. Any medical care associated with a diagnosis of cancer in the 183 days before and including the index date; a diagnosis of cancer for this purpose is any diagnostic code of International Classification of Diseases, 9th revision (ICD-9) in the range 140-208 "Malignant neoplasms …" or of the 10th revision (ICD-10) in the range C00-C96, "Malignant neoplasms"
2. Dispensing of methylnaltrexone for subcutaneous injection in the 183 days before and including the index date
3. Indication in the electronic records of the occurrence of MACE in the 183 days before and including the index date; see Section 9.3.2 "MACE" for screening criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients in this study will be 18 years of age or older, and they will have had at least 6 months of continuous data available before they enter one of the new-user cohorts. During the 6-month baseline period before cohort entry, they will have received at least 90 days of dispensed opioids, of which in the 60 days before cohort entry there were at least 30 days of opioids dispensed at an average of at least 30 morphine equivalent units (MEQ) per day. Patients will have no evidence of active cancer; they will have no evidence in the electronic record of MACE; they will not have received methylnatrexone bromide for subcutaneous injection. At the time of the index dispensing of naloxegol or comparison drug, cohort members will furthermore be current users of a dispensed opioid.
Sampling Method: Non-Probability Sample
Enrollment: 8800 (Estimated)
Dates: Start 2016-06-24 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiovascular events | can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 8 years
  while exposed to naloxegol or comparator exposure, composite of major adverse cardiovascular events which includes cardiovascular death, nonfatal myocardial infarction, and nonfatal stroke

CONTACTS AND LOCATIONS:
Overall Officials: Beth Nordstrom, Principal Investigator — Evidera
Locations (2):
- United States (2):
  - Research Site, Wilmington, Delaware
  - Research Site, Hines, Illinois